CLINICAL TRIAL: NCT06269081
Title: Testing the Efficacy of Two Interventions to Improve Health Outcomes and Quality of Life Among Rural Older Adults Living With HIV
Brief Title: Testing Two Interventions to Improve Health Outcomes and Quality of Life Among Rural Older Adults Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jennifer Walsh, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01NR020770 (NIH); R01NR020770 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Supportive-Expressive Peer Social Support Group + Individual Strengths-Based Case Management (Experimental)
  Interventions: Behavioral: Supportive-Expressive Peer Social Support Group Intervention; Behavioral: Individual Strengths-Based Case Management Intervention
- Supportive-Expressive Peer Social Support Group (Experimental)
  Interventions: Behavioral: Supportive-Expressive Peer Social Support Group Intervention
- Individual Strengths-Based Case Management (Experimental)
  Interventions: Behavioral: Individual Strengths-Based Case Management Intervention
- HIV Information Only (No Intervention): This arm will not receive either of the interventions but will receive information on successfully aging with HIV.

INTERVENTIONS:
Behavioral: Supportive-Expressive Peer Social Support Group Intervention — The social support group intervention involves weekly virtual support group meetings for 8 consecutive weeks. The groups, facilitated by trained research staff, will last approximately 90 minutes each week and include 5-12 individuals per group. Groups will follow pre-determined topic areas, with participants encouraged to explore their feelings about the difficulties associated with normal aging, being HIV-positive, and living with HIV/AIDS as an older adult. Facilitators will encourage mutual support among group members, promote greater openness and emotional expressiveness, and help participants to improve their social and family support and enhance their quality of life. This intervention is an adaptation of Telephone Supportive-Expressive Group Therapy.
  Arms: Supportive-Expressive Peer Social Support Group; Supportive-Expressive Peer Social Support Group + Individual Strengths-Based Case Management
Behavioral: Individual Strengths-Based Case Management Intervention — The strengths-based case management (SBCM) intervention helps participants address the multiple structural barriers faced by rural older people living with HIV. This intervention, delivered by trained research staff, includes two 60-minute telephone- or video-based SBCM counseling sessions, with shorter follow-up sessions to check-in on progress and help patients navigate identified barriers. The case manager will provide tailored sessions based on individually-identified needs and proximal life stressors. Capitalizing on participants' personal strengths, case managers will help empower participants to navigate issues related to employment, insurance, mental health, housing, or transportation. This may include assistance understanding, applying for, and accessing benefits or programs.
  Arms: Individual Strengths-Based Case Management; Supportive-Expressive Peer Social Support Group + Individual Strengths-Based Case Management

SUMMARY:
Engagement in HIV medical care and adherence to HIV medications are both essential in improving health outcomes among people living with HIV (PLH), but PLH living in rural areas-who suffer higher mortality rates than their urban counterparts-can confront multiple barriers to care engagement and adherence, especially as they face the logistical, medical, and social challenges associated with aging. This project will test the efficacy of two interventions to determine their impact on HIV health outcomes and quality of life among rural, older PLH living in the Southern U.S. The two interventions, adapted from evidence-based interventions and delivered remotely, are: (1) supportive-expressive peer social support groups and (2) strengths-based case management. We hypothesize that both interventions will increase viral suppression, antiretroviral therapy adherence, and health-related quality of life and decrease depressive symptoms. Results from this study will provide us with tools to improve health outcomes for rural older people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or greater
* Living in a county with a score of .4 or higher on the index of relative rurality (IRR)
* Living in Alabama, Arkansas, Delaware, Florida, Georgia, Kentucky, Louisiana, Maryland, Mississippi, Missouri, North Carolina, Oklahoma, South Carolina, Tennessee, Texas, Virginia, or West Virginia
* Living with HIV
* Has a telephone at home
* Able to provide informed consent

Exclusion Criteria:

* Not meeting eligibility criteria described above

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression | 4 and 12 month follow-ups
  HIV viral load will be assessed using self-collected dried blood spot (DBS) samples, with samples collecting using HemaSpot devices. Viral suppression will be defined as a measured viral load less than or equal to 839 copies/mL.
Antiretroviral Treatment Medication Adherence | 4, 8, and 12 month follow-ups
  Recent (past 30 day) antiretroviral treatment adherence will be self-reported using the 3-item Wilson Medication Adherence Scale. The calculated scale range is 0-100, with higher scores indicating more consistent medication adherence.
Health-Related Quality of Life | 4, 8, and 12 month follow-ups
  Health-related quality of life will be self-reported using the 31-item World Health Organization Quality of Life Brief Assessment for PLH (WHOQOL-HIV BREF). The calculated scale range is 0-100, with higher scores indicating better quality of life. Composite scores will be calculated in line with Walsh et al., 2024.
Depressive Symptoms | 4, 8, and 12 month follow-ups
  Depressive symptoms during the past 2 weeks will be self-reported via completion of the 9-item Patient Health Questionnaire-9 (PHQ-9). The calculated scale range is 0-27, with higher scores indicating more depressive symptoms.

SECONDARY OUTCOMES:
Social Support | 4, 8, and 12 month follow-ups
  Social support will be self-reported using the 19-item Medical Outcomes Study (MOS) Social Support Scale. Scale scores range from 1-5, with higher scores indicating more social support.
Loneliness | 4, 8, and 12 month follow-ups
  Loneliness will be self-reported using the 5-item Loneliness survey from the National Institutes of Health (NIH) Toolbox. Scale scores range from 1-5, with higher scores indicating greater loneliness.
Internalized HIV Stigma | 4, 8, and 12 month follow-ups
  Internalized HIV stigma will be self-reported using the 6-item internalized stigma subscale of the HIV Stigma Mechanisms scale. Scale scores range from 1-5, with higher scores indicating more internalized stigma.
General Self-Efficacy | 4, 8, and 12 month follow-ups
  General self-efficacy will be self-reported using the 8-item New General Self-Efficacy Scale. Scale scores range from 1-5, with higher scores indicating greater self-efficacy.
HIV Treatment Adherence Self-Efficacy | 4, 8, and 12 month follow-ups
  HIV treatment adherence self-efficacy will be self-reported using the 8-item HIV Treatment Adherence Self-Efficacy Scale (HIV-ASES). Scale scores range from 0-4, with higher scores indicating greater self-efficacy.
Accessing Needed Social and Medical Services | 4, 8, and 12 month follow-ups
  Participants will self-report which of 12 HIV-related social and medical services they have needed during the previous 3 months, and which of these needed services they were able to obtain. A composite variable will indicate whether participants successfully accessed at least one needed service (0 = no, 1 = yes).
Structural Barriers | 4, 8, and 12 month follow-ups
  Participants will self-report structural barriers they have faced in the past 3 months, with items assessing the following barriers: not having current health insurance, transportation as a barrier to health care, finances as a barrier to health care, not having enough food to eat, not having stable housing, and lacking eHealth literacy. Participants will be coded as having faced or not having faced each barrier, and barriers will be summed to indicate a score from 0-6, with higher scores indicating more structural barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Walsh, PhD, Principal Investigator — Center for AIDS Intervention Research, Medical College of Wisconsin; Andrew Petroll, MD, Principal Investigator — Center for AIDS Intervention Research, Medical College of Wisconsin
Locations (1):
- Center for AIDS Intervention Research, Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] O'Connell KA, Skevington SM. An international quality of life instrument to assess wellbeing in adults who are HIV-positive: a short form of the WHOQOL-HIV (31 items). AIDS Behav. 2012 Feb;16(2):452-60. doi: 10.1007/s10461-010-9863-0. PMID 21181253
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Earnshaw VA, Smith LR, Chaudoir SR, Amico KR, Copenhaver MM. HIV stigma mechanisms and well-being among PLWH: a test of the HIV stigma framework. AIDS Behav. 2013 Jun;17(5):1785-95. doi: 10.1007/s10461-013-0437-9. PMID 23456594
- [Background] Salsman JM, Butt Z, Pilkonis PA, Cyranowski JM, Zill N, Hendrie HC, Kupst MJ, Kelly MA, Bode RK, Choi SW, Lai JS, Griffith JW, Stoney CM, Brouwers P, Knox SS, Cella D. Emotion assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S76-86. doi: 10.1212/WNL.0b013e3182872e11. PMID 23479549
- [Background] Kidder DP, Wolitski RJ, Campsmith ML, Nakamura GV. Health status, health care use, medication use, and medication adherence among homeless and housed people living with HIV/AIDS. Am J Public Health. 2007 Dec;97(12):2238-45. doi: 10.2105/AJPH.2006.090209. Epub 2007 Oct 30. PMID 17971562
- [Background] Johnson MO, Neilands TB, Dilworth SE, Morin SF, Remien RH, Chesney MA. The role of self-efficacy in HIV treatment adherence: validation of the HIV Treatment Adherence Self-Efficacy Scale (HIV-ASES). J Behav Med. 2007 Oct;30(5):359-70. doi: 10.1007/s10865-007-9118-3. Epub 2007 Jun 23. PMID 17588200
- [Background] Chen, G., Gully, S. M., & Eden, D. (2001). Validation of a new general self-efficacy scale. Organizational research methods, 4, 62-83.
- [Background] Heckman TG, Heckman BD, Anderson T, Lovejoy TI, Mohr D, Sutton M, Bianco JA, Gau JT. Supportive-expressive and coping group teletherapies for HIV-infected older adults: a randomized clinical trial. AIDS Behav. 2013 Nov;17(9):3034-44. doi: 10.1007/s10461-013-0441-0. PMID 23474642
- [Derived] Petroll AE, Hirshfield S, Quinn KG, John SA, Algiers OH, Randall L, Wyley Long D, McAuliffe T, Walsh JL. Testing the Efficacy of 2 Interventions to Improve Health Outcomes and Quality of Life Among Rural Older Adults Living With HIV: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 17;14:e71429. doi: 10.2196/71429. PMID 41105943